CLINICAL TRIAL: NCT03424187
Title: The Acute Effects of Food Structure on Post Prandial Glucose and Subsequent Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 15HH3069
Record Dates: First submitted 2017-09-01; First posted 2018-02-06 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cicerin protein, Cicer arietinum

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- whole chickpea (Experimental): a test meal containing 26g available carbohydrates from chickpea (full structure)
  Interventions: Dietary Supplement: chickpea
- flour chickpea (Experimental): a test meal containing 26g available carbohydrates from flour chickpea (destroyed structure)
  Interventions: Dietary Supplement: chickpea
- intact cell chickpea (Experimental): a test meal containing 26g available carbohydrates from intact cell chickpea flour (full structure)
  Interventions: Dietary Supplement: chickpea

INTERVENTIONS:
Dietary Supplement: chickpea — all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea

SUMMARY:
Aims: To investigate the effects of different food structures on glucose concentrations and subsequent metabolic responses including insulin,GIP, GLP-1 DESIGN: A randomised, controlled, clinical trial.

DETAILED DESCRIPTION:
Rationale:

There is very little evidence at the present time in the role of food structure in glucose homeostasis. There is circumstantial evidence that foods consumed intact have great effects on suppressing appetite.

To test the effect of three structurally different meals with the same nutritional content and volume on appetite regulation. Each participant will receive the following meals:

Solid meal group. Milled (intact-cell) meal group. Milled (destroyed-cell) meal group.

All of which will contain the same macro and micro nutrients from the same food sources

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female
* Age ≥ 18 years ≤ 65 years
* Normal weight as classified by BMI 20-29.9 kg/m2
* Healthy, not diagnosed with any chronic diseases assessed as appropriate for inclusion, based on the pre-study screening.
* Willingness and ability to understand, participate and to comply with the study requirements
* Willingness and ability to give written informed consent

Exclusion Criteria:

* Has thyroid defects
* Under hormone or steroids therapy
* Is pregnant or lactating (female)
* Had given birth within the past year (female)
* Is taking drugs that could affect appetite or plasma glucose levels.
* Is taking natural remedies that modulate appetite or plasma glucose levels.
* Has excessive alcohol intake
* Had blood donation within 12wks prior to start date
* Psychiatric illness
* Smokers
* History of any disease with unknown outcome
* Has diabetes
* Has nut allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-07 (Actual)

REFERENCES:
- [Derived] Alshaalan RA, Charalambides MN, Edwards CH, Ellis PR, Alrabeah SH, Frost GS. Impact of chickpea hummus on postprandial blood glucose, insulin and gut hormones in healthy humans combined with mechanistic studies of food structure, rheology and digestion kinetics. Food Res Int. 2024 Jul;188:114517. doi: 10.1016/j.foodres.2024.114517. Epub 2024 May 10. PMID 38823849

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: this study was a randomized crossover study
Groups:
- Experimental: Whole Chickpea First, Then Flour Chickpea, Then Intact Cell Chickpea: First intervention whole chickpea hummus (26g carbohydrate), washout (1 week), Second Flour chickpea hummus (26g carbohydrate), washout (1 week), Third Intact Cell Chickpea hummus (26g carbohydrate)
- Experimental: Whole Chickpea First, Then Intact Cell Chickpea, Then Flour Chickpea: First intervention whole chickpea hummus (26g carbohydrate), washout (1 week), Second Intact Cell Chickpea hummus (26g carbohydrate), washout (1 week), Third Flour chickpea hummus (26g carbohydrate)
- Experimental:Flour Chickpea First, Then Whole Chickpea, Then Intact Chickpea: First intervention Flour chickpea hummus (26g carbohydrate), washout (1 week), Second whole Chickpea hummus (26g carbohydrate), washout (1 week), Third Intact Cell hummus (26g carbohydrate)
- Experimental: Flour Chickpea First, Intact Cell Chickpea, Whole Chickpea: First intervention Flour chickpea hummus (26g carbohydrate), washout (1 week), Second Intact Cell Chickpea hummus (26g carbohydrate), washout (1 week), Third whole chickpea hummus (26g carbohydrate)
- Experimental: Intact Cell Chickpea First, Then Whole Chickpea, Then Flour Chickpea: First intervention Intact Cell hummus (26g carbohydrate), washout (1 week), Second whole Chickpea hummus (26g carbohydrate), washout (1 week), Third Flour chickpea hummus (26g carbohydrate)
- Experimental: Intact Cell Chickpea First, Then Flour Chickpea, Then Whole Chickpea: First intervention Intact Cell hummus (26g carbohydrate), washout (1 week), Second flour Chickpea hummus (26g carbohydrate), washout (1 week), Third whole chickpea hummus (26g carbohydrate)
Period: Overall Study
Arm/Group | Experimental: Whole Chickpea First, Then Flour Chickpea, Then Intact Cell Chickpea | Experimental: Whole Chickpea First, Then Intact Cell Chickpea, Then Flour Chickpea | Experimental:Flour Chickpea First, Then Whole Chickpea, Then Intact Chickpea | Experimental: Flour Chickpea First, Intact Cell Chickpea, Whole Chickpea | Experimental: Intact Cell Chickpea First, Then Whole Chickpea, Then Flour Chickpea | Experimental: Intact Cell Chickpea First, Then Flour Chickpea, Then Whole Chickpea
Started | 2 | 3 | 2 | 3 | 2 | 3
Completed | 2 | 3 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Whole Chickpea First, Then Intact Cell Chickpea, Then Flour Chickpea: First intervention whole chickpea hummus (26g carbohydrate), washout (1 week), Second Intact Cell Chickpea hummus (26g carbohydrate), washout (1 week), Third Flour chickpea hummus (26g carbohydrate
- Total: Total of all reporting groups
Arm/Group | Experimental: Whole Chickpea First, Then Flour Chickpea, Then Intact Cell Chickpea | Experimental: Whole Chickpea First, Then Intact Cell Chickpea, Then Flour Chickpea | Experimental:Flour Chickpea First, Then Whole Chickpea, Then Intact Chickpea | Experimental: Flour Chickpea First, Intact Cell Chickpea, Whole Chickpea | Experimental: Intact Cell Chickpea First, Then Whole Chickpea, Then Flour Chickpea | Experimental: Intact Cell Chickpea First, Then Flour Chickpea, Then Whole Chickpea | Total
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 3 | 2 | 3 | 15
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 2 | 1 | 10
  Male | 0 | 0 | 1 | 2 | 0 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-prandial Glucose Concentrations
Description: Blood glucose concentrations were assessed for each participant after each test meal: whole chickpea hummus, Flour chickpea hummus, and Intact cell chickpea hummus. Blood samples were collected before the introduction of the test meal and then at 15 minutes, 30 min, 60, 90, 120, and 180 minutes after the consumption of the test meal.
  Data were not collected for intact cell chickpea hummus
Time Frame: before the consumption of the test meal and then 15 min, 30, 60,90, 120, 180 minutes after the consumption of the test meal.
Population: Blood glucose concentrations were assessed for each participant after each test meal: whole chickpea hummus, Flour chickpea hummus only. Blood samples were collected before the introduction of the test meal and then at 15 minutes, 30 min, 60, 90, 120, and 180 minutes after the consumption of the test meal.
Measure: Mean (Standard Deviation); unit: mmol/l
Groups:
- Whole Chickpea: a test meal containing 26g available carbohydrates from chickpea (full structure)
  chickpea: all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea
- Flour Chickpea: a test meal containing 26g available carbohydrates from flour chickpea (destroyed structure)
  chickpea: all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea
Arm/Group | Whole Chickpea | Flour Chickpea
Number analyzed (Participants) | 15 | 15
mmol/l
  time point 0 | 4.9 (0.48) | 4.8 (0.31)
  Time point 15 | 4.9 (0.53) | 5.01 (0.38)
  Time point 30 | 5.1 (0.57) | 5.4 (0.53)
  Time point 60 | 5.08 (0.78) | 4.9 (0.87)
  Time point 90 | 5.07 (0.73) | 4.8 (0.6)
  Time point 120 | 5.18 (0.56) | 4.9 (0.4)
  Time point 180 | 5.14 (0.46) | 5.1 (0.44)

2. Primary Outcome: Post-prandial Blood Insulin Concentrations
Description: Blood glucose concentrations were assessed for each participant after each test meal: whole chickpea hummus, Flour chickpea hummus, and Intact cell chickpea hummus. Blood samples were collected before the introduction of the test meal and then at 15 minutes, 30 min, 60, 90, 120, and 180 minutes after the consumption of the test meal.
Time Frame: before the consumption of the test meal and then 15, 30, 60, 90, 120, and 180 minutes post consumption of test meal.
Measure: Mean (Standard Deviation); unit: uU/ml
Groups:
- Whole Chickpea Hummus: a test meal containing 26g available carbohydrates from chickpea (full structure)
  chickpea: all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea
- Flour Chickpea Hummus: a test meal containing 26g available carbohydrates from flour chickpea (destroyed structure)
  chickpea: all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea
- Intact Cell Chickpea Hummus: a test meal containing 26g available carbohydrates from intact cell chickpea flour (full structure)
  chickpea: all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea
Arm/Group | Whole Chickpea Hummus | Flour Chickpea Hummus | Intact Cell Chickpea Hummus
Number analyzed (Participants) | 15 | 15 | 15
uU/ml
  0 minutes | 9.3 (4.03) | 10.3 (5.4) | 8.8 (5.4)
  15 minutes | 16.8 (9.6) | 20 (10.9) | 26.24 (19.6)
  30 minutes | 29.3 (12.5) | 37.5 (17.3) | 43.1 (26)
  60 minutes | 29.1 (20.4) | 36.5 (24.2) | 37.9 (23.2)
  90 minutes | 24.3 (15.8) | 31.6 (17.12) | 33.7 (13.8)
  120 minutes | 12.4 (14.2) | 34.1 (24.5) | 36.5 (31.1)
  180 minutes | 14.9 (8.5) | 16.8 (7.4) | 17.57 (7.7)

3. Secondary Outcome: Post-prandial Gut Hormone Gastric Inhibitory Polypeptide (GIP)
Description: Blood GIP concentrations were assessed for each participant after each test meal: whole chickpea hummus, and Flour chickpea hummus. Blood samples were collected before the introduction of the test meal and then at 15 minutes, 30 min, 60, 90, 120, and 180 minutes after the consumption of the test meal.
  Data were not collected for intact cell chickpea hummus
Time Frame: before the consumption of the test meal at 0 min and then post test meal at 15, 30,60 ,90,120 and 180 minutes.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Whole Chickpea Hummus | Flour Chickpea Hummus
Number analyzed (Participants) | 15 | 15
pmol/L
  baseline 0 minutes | 43.02 (23.07) | 47 (20.6)
  15 min | 102.6 (34.47) | 181.3 (97.3)
  30 min | 343.7 (166.9) | 516.2 (217.9)
  60 min | 508 (186.8) | 651 (220)
  90 min | 509 (199.5) | 601.9 (199)
  120 min | 466.48 (171.32) | 562.033 (172.6)
  180 min | 378.1 (153.9) | 440.7 (199.4)

4. Secondary Outcome: Post-prandial Gut Hormone Glucagon-like Peptide 1 (GLP-1)
Description: Blood GLP-1 concentrations were assessed for each participant after each test meal: whole chickpea hummus, Flour chickpea hummus, and Intact cell chickpea hummus. Blood samples were collected before the introduction of the test meal and then at 15 minutes, 30 min, 60, 90, 120, and 180 minutes after the consumption of the test meal.
Time Frame: baseline before the consumption of the test meal, and then 15,30,60,90,120,180 min after the consumption of the test meal.
Measure: Mean (Standard Deviation); unit: pmol/l
Groups:
- Whole Chickpea Hummus: a test meal containing 26g available carbohydrates from chickpea (full structure)
- Flour Chickpea Hummus: a test meal containing 26g available carbohydrates from flour chickpea (destroyed structure)
- Intact Cell Chickpea Hummus: a test meal containing 26g available carbohydrates from Intact cell chickpea (destroyed structure)
Arm/Group | Whole Chickpea Hummus | Flour Chickpea Hummus | Intact Cell Chickpea Hummus
Number analyzed (Participants) | 15 | 15 | 15
pmol/l
  baseline | 67.3 (27.1) | 85.3 (36.5) | 80.8 (31.2)
  15 min | 122.8 (63.3) | 98.7 (49.3) | 91.7 (34.2)
  30 min | 108.8 (59.5) | 110.7 (33) | 123.2 (45.8)
  60 min | 113.5 (39.4) | 115.5 (43.2) | 128 (42)
  90 min | 134.5 (65.7) | 119 (37.5) | 120.3 (66.5)
  120 min | 114.6 (77) | 130.9 (57.6) | 108 (46.4)
  180 min | 103.9 (57.7) | 109.2 (53) | 92.9 (49.4)

5. Secondary Outcome: Energy Intake at a Meal Given in Excess
Description: The difference in ad libitum food intake after 210 minutes post test meal to test the difference of energy intake following whole chickpea hummus, flour chickpea hummus, and intact cell chickpea hummus.
Time Frame: post consumption of the test meal at 120 minutes
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Whole Chickpea Hummus | Flour Chickpea Hummus | Intact Cell Chickpea Hummus
Number analyzed (Participants) | 15 | 15 | 15
Kcal | 628.03 (321.7) | 681.9 (326) | 724.7 (308.3)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Intact Cell Chickpea: a test meal containing 26g available carbohydrates from intact cell chickpea flour (full structure)
  chickpea: all three meals are isocaloric but different in the chickpea structure( physical form):
  • Whole chickpea, flour chickpea, intact cell flour chickpea
Arm/Group | Whole Chickpea | Flour Chickpea | Intact Cell Chickpea
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT03424187/SAP_000.pdf
  • Study Protocol (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT03424187/Prot_001.pdf